CLINICAL TRIAL: NCT06053489
Title: Effect of Remimazolam and Sevoflurane Anesthesia on Recovery in Pediatric Patients Who Underwent Ophthalmic Surgery Under General Anesthesia
Brief Title: Effect of Remimazolam and Sevoflurane Anesthesia on Recovery in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant professor for fund, Pusan National University Yangsan Hospital
Other Study IDs: 2023-09-09
Record Dates: First submitted 2023-09-09; First posted 2023-09-25 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Ophthalmic Abnormalities; Pediatric Disorder
MeSH Terms: interventions — Anesthesia, General; remimazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: general anesthesia with remimazolam — general anesthesia with remimazolam in pediatric patients undergoing ophthalmic surgery

SUMMARY:
The most commonly used anesthetic for general anesthesia in pediatric patients is sevoflurane, an inhalation anesthetic. However, the incidence of emergence agitation after sevoflurane anesthesia in pediatric patients is high, with reports of up to 67%. Remimazolam (Byfavo Inj., Hana Pharm Col, Ltd., Seoul, Korea) has a short context-sensitive half-life of 7.5 minutes, and the time it takes from the end of anesthesia until the patient wakes up is predictable. According to a study by Yang X et al., administering a small amount of remimazolam (0.2 mg/kg) intravenously at the end of general anesthesia using sevoflurane reduced the incidence of emergence agitation. However, very few studies have evaluated the use of remimazolam in general anesthesia in pediatric patients.

DETAILED DESCRIPTION:
* The most commonly used anesthetic for general anesthesia in pediatric patients is sevoflurane, an inhalation anesthetic. It has the advantage of being able to induce anesthesia without securing an intravenous route and causing less irritation to the airway. However, the incidence of emergence agitation after sevoflurane anesthesia in pediatric patients is high, with reports of up to 67%. Emergence agitation can cause physical damage to the patient, workload in the recovery room, and dissatisfaction of the caregiver.
* Remimazolam (Byfavo Inj., Hana Pharm Col, Ltd., Seoul, Korea) is a benzodiazepine drug used for inducing and maintaining general anesthesia and for sedation during procedures. When remimazolam is used as a general anesthetic, it has the advantage of being metabolized quickly by enzymes in the liver compared to propofol, has a short context-sensitive half-life of 7.5 minutes, and can be reversed with flumazenil. Therefore, during general anesthesia using remimazolam, the time it takes from the end of anesthesia until the patient wakes up is predictable. According to a study by Yang X et al., administering a small amount of remimazolam (0.2 mg/kg) intravenously at the end of general anesthesia using sevoflurane reduced the incidence of emergence agitation.
* However, very few studies have evaluated the use of remimazolam in general anesthesia in pediatric patients and its effect on endotracheal extubation time after anesthesia in operating room, emergence agitation, pain, and discharge time in the postanesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 3 and 18 years old who underwent ophthalmic surgery under general anesthesia
* When anesthesia was induced and maintained with remimazolam, or anesthesia was induced with propofol and maintained with sevoflurane.

Exclusion Criteria:

- none

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged between 3 and 18 years old who underwent ophthalmic surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Time to extubation | Immediate after the end of general anesthesia
  Time to extubation after the end of general anesthesia

SECONDARY OUTCOMES:
Time for post-anesthesia recovery | From the time of immediate after entering the PACU until until achieving post-anesthesia recovery score of 9 or more, assessed up to 4 hours
  Time taken until the patient can leave the PACU. The post-anesthesia recovery score (modified Aldrete score) is used for assessment of patient's activity, respiration, blood pressure, consciousness, and peripheral oxygen saturation. A score 9 points or more is required for discharge from the PACU.
Postoperative pain | Immediate after entering the PACU, 15 minutes after entering the PACU
  Visual analog scale (VAS) is going to be measured after entering the PACU. The VAS is a validated, subjective measure for acute and chronic pain. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Incidence of emergence delirium | Immediate after entering the PACU, 15 minutes after entering the PACU
  Emergence delirium measured after entering the PACU
Adverse events and complications | during general anesthesia, and recovery after general anesthesia, up to 1 day
  Adverse events and complications that occur during anesthesia and recovery from anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital, Yangsan, South Korea
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No